CLINICAL TRIAL: NCT02779036
Title: The Effects of a Structured, Progressive, Task-oriented Home Exercise Program on Walking Competency in Individual Post Stroke
Brief Title: Optimizing Walking Function of Stroke Survivors by a Task-Oriented Home Exercise Program
Acronym: TOHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: University of Medical Technology, Yangon (Other); National Rehabilitation Hospital, Myanmar (Unknown); Yangon General Hospital, Myanmar (Unknown)
Responsible Party: Principal Investigator, Thin Thin Moe, Ph D candidate, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2016
Record Dates: First submitted 2016-05-15; First posted 2016-05-20 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2016-10

CONDITIONS: Stroke
Keywords: Stroke; task-oriented home exercise; walking competency; Usual Physiotherapy care
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Task-oriented Exercise (Experimental): Structured, progressive, task-oriented, home exercise program
  Interventions: Procedure: Task-oriented home exercise
- Usual Care (Active Comparator): Usual Physiotherapy Care
  Interventions: Procedure: Usual Physiotherapy Care

INTERVENTIONS:
Procedure: Task-oriented home exercise — Structured, walking related task-oriented home exercise program with three progressive steps, at moderate to high intensity, 60 minutes per session, three sessions per week for total 8 weeks.
  Arms: Task-oriented Exercise
Procedure: Usual Physiotherapy Care — Deficits-oriented free active and resisted lower extremity exercises with bicycling and overground walking , 60 minutes per session, three sessions per week for total 8 weeks.
  Arms: Usual Care

SUMMARY:
In a randomized-controlled study, the effects of a structured, progressive, task-oriented home exercise program to optimize walking competency will be evaluated in subacute stroke survivors.

DETAILED DESCRIPTION:
The majority of stroke individuals unable to reenter their previous community life after they have had a stroke. Reintegration of community life by optimizing walking function is a major goal of stroke rehabilitation. Because not widely available inpatient rehabilitation, discharged with incomplete recovery, limited numbers of technically trained physical therapists, financial saving, and transportation difficulty, home-based stroke rehabilitation setting has been interested in many developing countries.

Task- oriented exercise is well known and accepted approach to optimize walking function with underlying principles of motor control and motor learning theories. This approach has been used in the clinical setting with close supervision, but identification of appropriate protocol in the community environment is on progress. To date, no proper home exercise program based on task-oriental principle with minimal supervision for improving walking competency after stroke has been proposed in stroke rehabilitation.

The purpose of this study is to investigate the effects of a structured, progressive, task- oriented home exercise program on walking competency in individual post stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Either side of both type first stroke within 2 weeks to six months of onset with confirmatory diagnosis by CT Scan and MRI.
2. Age between 40 to 65 years old.
3. Moderate severity of stroke measured by the modified Rankin Scale (mRS- 3)
4. Able to comprehend the instructions with good cognition measured by Mini-Mental State Examination (MMSE > 23).
5. Postadoption stage of readiness to change measured by the Stages of Change Questionnaire (stage 4 and 5)

Exclusion Criteria:

1. Diagnosed with other neurological disorder such as Parkinson's disease, peripheral nerve injury.
2. Serious cardiac conditions (angina and myocardial infarction during the previous month, resting heart rate of more than 120, a systolic blood pressure of more than 180 mm Hg, and a diastolic blood pressure of more than 100 mm Hg)
3. Fugl Meyer Assessment score (lower extremity) less than ≤ 21
4. Significant hip, knee and ankle contracture that would limit ambulation (Fugl Meyer (ROM) ≤1 in each joint).
5. Orthopedic and rheumatological disorder with weight bearing pain (Fugl Meyer (pain) ≤ 1 in hip, knee and ankle joint movement).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
6 Minutes Walk Test | up to 8 weeks
  Patients will be measured their walking distance by a blind assessor on five occasions:at baseline,1,2,5 and 8 weeks after baseline testing.
10 Meter Walk Test | up to 8 weeks
  Patients will be measured their walking speed by a blind assessor on five occasions:at baseline,1,2,5 and 8 weeks after baseline testing.

SECONDARY OUTCOMES:
Berg Balance Scale | up to 8 weeks
  Patients will be measured their walking balance by a blind assessor on five occasions:at baseline,1,2,5 and 8 weeks after baseline testing.
Dynamic Gait Index | Baseline and 8 weeks
  Patients will be measured their walking adaptability by a blind assessor on two occasions:at baseline and 8 weeks after baseline testing.
Stroke Impact Scale (Participation) | Baseline and 8 weeks
  Patients will be measured their community participation by a blind assessor on two occasions:at baseline and 8 weeks after baseline testing.

CONTACTS AND LOCATIONS:
Overall Officials: Thin Thin Moe, M.Med.Tech, Principal Investigator — Mahidol University; Chutima Jalayondeja, Dr.P.H. MSc, Study Chair — Mahidol University; Sopa Pichaiyongwongdee, M.Sc. B.Sc, Study Director — Mahidol University; Vimonwan Hiengkaew, PhD. MSc, Study Director — Mahidol University; Jarugool Tretriluxana, PhD. MSc, Study Director — Mahidol University
Locations (2):
- Burma (2):
  - National Rehabilitation Hospital, Yangon
  - Physical Medicine and Rehabilitation Department, Yangon General Hospital, Yangon

IPD SHARING:
Plan to Share IPD: Undecided